CLINICAL TRIAL: NCT06510647
Title: Risk Factors for Hormonal Therapy Failure in Patients With Endometriosis.
Acronym: ENDOFAIL-01
Status: Recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Full Professor of Gynecology and Obstetrics, University of Cagliari
Other Study IDs: ENDOFAIL-01
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Endometriosis
Keywords: endometriosis; hormonal therapy; risk factors; therapy failure
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients with endometriosis who are non-responsive to medical therapy after 12 months
  Interventions: Other: Hormonal Therapy Agent
- Group B: Patients with endometriosis who are responsive to medical therapy after 12 months
  Interventions: Other: Hormonal Therapy Agent

INTERVENTIONS:
Other: Hormonal Therapy Agent — With an endometriosis diagnosis in which hormonal therapy is indicated, patients who satisfy inclusion and exclusion criteria will be administered scientifically validated questionnaires at the time of the visit (time 0): Endometriosis Health Profile-30 and the Short Form Health Survey SF-12.
  The second evaluation will be conducted 6 months later (time 1) along with a gynecological examination and gynecological ultrasound, and the same two questionnaires will be administered. Patients will be defined as non-responsive to medical therapy if their Endometriosis Health Profile 30 scores are equal to or higher at the "time 1" visit compared to the enrollment visit at "time 0".
  Patients will then be re-evaluated 12 months (time 2) after the first visit with the same criteria, and the two questionnaires will be administered once more. Similarly, patients with EHP-30 scores equal to or higher than the previous control at time 1 will be defined as non-responsive to medical therapy.

SUMMARY:
The primary objective of our study is to determine the percentage of patients with endometriosis who are non-responsive to medical therapy after 12 months and to compare the clinical and ultrasound characteristics of this group of patients (study group) with the clinical and ultrasound characteristics of patients who are responsive to medical therapy (control group).

The secondary objective of the study will be to determine the percentage of patients with endometriosis who are non-responsive to medical therapy after 6 months and to compare the clinical and ultrasound characteristics of this group of patients (study group) with the clinical and ultrasound characteristics of patients who are responsive to medical therapy (control group).

DETAILED DESCRIPTION:
This will be an observational study without the use of medication, multicentric, prospective.

Patients aged between 18 and 50 years, with a clinical and ultrasound diagnosis of endometriosis painful symptoms related to endometriosis (dyspareunia, dyschezia, dysmenorrhea, chronic pelvic pain, dysuria, periovulatory pain, with at least one of these symptoms presenting a Numerical Pain Rating Scale intensity > 5), with an indication for hormonal therapy will be included after the acquisition of informed consent.

On the other hand, patients with contraindications to oral hormonal therapy, those with current or past pelvic infections, with a history of malignancy or current suspicion of malignant gynecological lesions, previous pelvic surgery (hysterectomy, salpingectomy, ovarian cyst removal, myomectomy, surgery for endometriosis, intestinal resections), positive history for other causes of chronic pelvic pain, or women in postmenopausal status will be excluded.

Enrollment will take place among patients who access the specialized endometriosis clinics of the Department of Gynecology and Obstetrics - Prof. Stefano Angioni, and participating centers for an initial visit. During this visit, as per clinical practice, a gynecological examination and a transvaginal gynecological ultrasound will be performed by an expert operator. In the case of an endometriosis diagnosis for which hormonal therapy is indicated and the inclusion and exclusion criteria are met, the patient will be asked to sign the informed consent for participation in the study and consent to the processing of personal data. These patients will be administered scientifically validated questionnaires at the time of the visit (time 0): Endometriosis Health Profile - 30 and the Short Form Health Survey SF - 12 ). The first is a questionnaire widely used in studies analyzing the quality of life of patients with endometriosis as it is specific to the disease, while the second is a generic quality of life questionnaire widely used in literature.

The second evaluation will be conducted 6 months later (time 1) along with a gynecological examination and gynecological ultrasound as per the normal care pathway, and the same questionnaires administered during the enrollment visit will be given again. Patients will be defined as non-responsive to medical therapy if their Endometriosis Health Profile 30 scores are equal to or higher at the "time 1" visit compared to the enrollment visit at "time 0".

Patients will then be re-evaluated, as per normal clinical practice, 12 months (time 2) after the first visit, again through a gynecological examination and gynecological ultrasound, and the two aforementioned questionnaires will be administered once more. Similarly, patients with EHP-30 scores equal to or higher than the previous control at time 1 will be defined as non-responsive to medical therapy.

The study will be discontinued for patients who, at the first follow-up visit, show EHP-30 scores lower than the previous control (therefore considered responsive) but who request to discontinue or switch therapy due to side effects deemed disabling. These patients will only be included in the analysis related to the 6-month outcome objective, their characteristics will be examined through descriptive analysis, and an attrition analysis with logistic regression will be conducted to identify variables potentially associated with dropping out of the study.

At Times 0, 1, and 2, the following parameters will be recorded:

* Age, BMI, parity, comorbidities, pain symptoms (endometriosis-related pain score), characteristics of bowel habits and urination, locations and characteristics of endometriotic lesions, type of hormonal therapy;
* Results of the administered questionnaires.

The total duration of the study will be 5 years and 7 months, divided as follows:

* Enrollment: 52 months
* Minimum follow-up: 12 months
* Data analysis: 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years;
* Patients with painful symptoms related to endometriosis (dyspareunia, dyschezia, dysmenorrhea, chronic pelvic pain, dysuria, periovulatory pain, with at least one of these symptoms presenting a Numerical Pain Rating Scale intensity > 5);
* Indication for the administration of oral hormonal medical therapy for endometriosis;
* Acquisition of informed consent.

Exclusion Criteria:

* Patients with contraindications to oral hormonal therapy;
* Current or past pelvic infections;
* History of malignancy or current suspicion of malignant gynecological lesions;
* Previous pelvic surgery (hysterectomy, salpingectomy, ovarian cyst removal, myomectomy, surgery for endometriosis, intestinal resections);
* Positive history for other causes of chronic pelvic pain;
* Postmenopausal status.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a clinical and ultrasound diagnosis of endometriosis with an indication for hormonal therapy.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with endometriosis who are non-responsive to medical therapy after 12 months | 12 months
  To determine the percentage of patients with endometriosis who are non-responsive to medical therapy after 12 months and to compare the clinical and ultrasound characteristics of this group of patients (study group) with the clinical and ultrasound characteristics of patients who are responsive to medical therapy (control group).

SECONDARY OUTCOMES:
Percentage of patients with endometriosis who are non-responsive to medical therapy after 6 months | 6 months
  To determine the percentage of patients with endometriosis who are non-responsive to medical therapy after 6 months and to compare the clinical and ultrasound characteristics of this group of patients (study group) with the clinical and ultrasound characteristics of patients who are responsive to medical therapy (control group).

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico "Duilio-Casula", Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dunselman GA, Vermeulen N, Becker C, Calhaz-Jorge C, D'Hooghe T, De Bie B, Heikinheimo O, Horne AW, Kiesel L, Nap A, Prentice A, Saridogan E, Soriano D, Nelen W; European Society of Human Reproduction and Embryology. ESHRE guideline: management of women with endometriosis. Hum Reprod. 2014 Mar;29(3):400-12. doi: 10.1093/humrep/det457. Epub 2014 Jan 15. PMID 24435778
- [Background] Cornillie FJ, Oosterlynck D, Lauweryns JM, Koninckx PR. Deeply infiltrating pelvic endometriosis: histology and clinical significance. Fertil Steril. 1990 Jun;53(6):978-83. doi: 10.1016/s0015-0282(16)53570-5. PMID 2140994
- [Background] Montanari G, Di Donato N, Benfenati A, Giovanardi G, Zannoni L, Vicenzi C, Solfrini S, Mignemi G, Villa G, Mabrouk M, Schioppa C, Venturoli S, Seracchioli R. Women with deep infiltrating endometriosis: sexual satisfaction, desire, orgasm, and pelvic problem interference with sex. J Sex Med. 2013 Jun;10(6):1559-66. doi: 10.1111/jsm.12133. Epub 2013 Apr 3. PMID 23551753
- [Background] Seracchioli R, Poggioli G, Pierangeli F, Manuzzi L, Gualerzi B, Savelli L, Remorgida V, Mabrouk M, Venturoli S. Surgical outcome and long-term follow up after laparoscopic rectosigmoid resection in women with deep infiltrating endometriosis. BJOG. 2007 Jul;114(7):889-95. doi: 10.1111/j.1471-0528.2007.01363.x. Epub 2007 May 15. PMID 17501958
- [Background] Stratton P, Khachikyan I, Sinaii N, Ortiz R, Shah J. Association of chronic pelvic pain and endometriosis with signs of sensitization and myofascial pain. Obstet Gynecol. 2015 Mar;125(3):719-728. doi: 10.1097/AOG.0000000000000663. PMID 25730237
- [Background] Vercellini P, Buggio L, Somigliana E. Role of medical therapy in the management of deep rectovaginal endometriosis. Fertil Steril. 2017 Dec;108(6):913-930. doi: 10.1016/j.fertnstert.2017.08.038. PMID 29202965
- [Background] Becker CM, Gattrell WT, Gude K, Singh SS. Reevaluating response and failure of medical treatment of endometriosis: a systematic review. Fertil Steril. 2017 Jul;108(1):125-136. doi: 10.1016/j.fertnstert.2017.05.004. PMID 28668150
- [Background] Jones G, Kennedy S, Barnard A, Wong J, Jenkinson C. Development of an endometriosis quality-of-life instrument: The Endometriosis Health Profile-30. Obstet Gynecol. 2001 Aug;98(2):258-64. doi: 10.1016/s0029-7844(01)01433-8. PMID 11506842
- [Background] Del Forno S, Mabrouk M, Arena A, Mattioli G, Giaquinto I, Paradisi R, Seracchioli R. Dienogest or Norethindrone acetate for the treatment of ovarian endometriomas: Can we avoid surgery? Eur J Obstet Gynecol Reprod Biol. 2019 Jul;238:120-124. doi: 10.1016/j.ejogrb.2019.04.010. Epub 2019 May 2. PMID 31132690